CLINICAL TRIAL: NCT05279417
Title: Phase 2b, Randomized, Multicenter, Double-blind, Parallel Group, Placebo Controlled, Dose Ranging Study to Investigate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of ATI-450 Plus Methotrexate (MTX) Versus Placebo Plus MTX in Patients With Moderate to Severe Active Rheumatoid Arthritis (RA) Who Have Had an Inadequate Response to MTX Alone
Brief Title: ATI-450 Plus Methotrexate (MTX) Versus Placebo Plus MTX in Participants With Moderate to Severe Active Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATI-450-RA-202; 2021-002860-31 (EudraCT Number)
Record Dates: First submitted 2022-02-18; First posted 2022-03-15 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid; Arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATI-450 20 mg BID plus Methotrexate (Experimental): ATI-450 20 mg oral tablet twice daily (BID) with a stable weekly dose of methotrexate for 12 weeks
  Interventions: Drug: Methotrexate; Drug: ATI-450 20 mg oral tablet BID
- ATI-450 50 mg BID plus Methotrexate (Experimental): ATI-450 50 mg oral tablet BID with a stable weekly dose of methotrexate for 12 weeks
  Interventions: Drug: ATI-450 50 mg oral tablet BID; Drug: Methotrexate
- Placebo plus Methotrexate (Placebo Comparator): Placebo oral tablet BID with a stable weekly dose of methotrexate for 12 weeks
  Interventions: Drug: Placebo oral tablet; Drug: Methotrexate

INTERVENTIONS:
Drug: ATI-450 50 mg oral tablet BID — Oral, small molecule MK2 inhibitor
  Other Names: zunsemetinib
  Arms: ATI-450 50 mg BID plus Methotrexate
Drug: Placebo oral tablet — Placebo tablet manufactured to match ATI-450 in appearance
  Arms: Placebo plus Methotrexate
Drug: Methotrexate — 15 mg to 25 mg weekly
Drug: ATI-450 20 mg oral tablet BID — Oral, small molecule MK2 inhibitor
  Other Names: zunsemetinib
  Arms: ATI-450 20 mg BID plus Methotrexate

SUMMARY:
This study evaluates ATI-450 plus MTX versus placebo plus MTX in participants with moderate to severe active RA who have had an inadequate response to MTX alone.

DETAILED DESCRIPTION:
This is a Phase 2b, randomized, multicenter, double-blind, parallel group, placebo controlled, dose ranging study to investigate the efficacy, safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple doses of ATI-450 plus MTX versus placebo plus MTX in participants with moderate to severe active RA who have had an inadequate response to MTX alone.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and be willing to sign the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved participant ICF prior to administration of any study-related procedures.
* Diagnosis of adult-onset RA as defined by the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria.
* Have active moderate to severe RA at Screening.
* A minimum of 12 weeks on MTX with a stable MTX dose.

Exclusion Criteria:

* Current acute or chronic immunoinflammatory disease other than RA which may impact the course or assessment of RA.
* Uncontrolled non-immunoinflammatory disease that may place the participant at increased risk during the study or impact the interpretation of results (eg, previous malignancy, recurrent infection, previous venous thromboembolism).
* Participant has experience with > 2 biologics, > 1 JAK inhibitor, or a combination of 1 biologic experience and 1 JAK inhibitor.
* Currently receiving corticosteroids at doses > 10 mg/day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving ACR20 at Week 12 | Baseline to Week 12

SECONDARY OUTCOMES:
Proportion of patients achieving ACR50/70 at Week 12 | Baseline to Week 12
Proportion of patients achieving ACR20/50/70 over time | Up to 12 Weeks
Mean change from baseline in DAS28-CRP over time | Up to 12 Weeks
Proportion of patients achieving DAS28-CRP remission (score < 2.6) over time | Up to 12 Weeks
Proportion of patients achieving DAS28-CRP low disease activity (score ≤ 3.2) over time | Up to 12 Weeks
Mean change from baseline in CDAI over time | Up to 12 Weeks
Proportion of patients achieving CDAI remission (score ≤ 2.8) over time | Up to 12 Weeks
Percent change from baseline in hsCRP level over time | Up to 30 days after 12 weeks of treatment
Health Assessment Questionnaire-Disability Index (HAQ-DI) score over time | Up to 12 Weeks
Short Form Health Survey version-2.0 (SF-36v2) score over time | Up to 12 Weeks
Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) score over time | Up to 12 Weeks
Incidence of adverse events (AEs), serious AEs (SAEs), laboratory value abnormalities, electrocardiogram (ECG) abnormalities, vital signs abnormalities | Baseline to Week 12
Trough ATI-450 and metabolite (CDD-2164) concentrations at clinic visits (trough and 2-hour post dose will be collected). | Study Days 1, 8, and 85

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Aggarwal, Study Director — Aclaris Therapeutics, Inc.
Locations (41):
- United States (11):
  - Aclaris Investigational Site, El Cajon, California
  - Aclaris Investigational Site, Encino, California
  - Aclaris Investigational Site, La Jolla, California
  - Aclaris Investigational Site, Palm Desert, California
  - Aclaris Investigational Site, Tampa, Florida
  - Aclaris Investigational Site, Oklahoma City, Oklahoma
  - Aclaris Investigational Site, Duncansville, Pennsylvania
  - Aclaris Investigational Site, Jackson, Tennessee
  - Aclaris Investigational Site, Cypress, Texas
  - Aclaris Investigational Site, Mesquite, Texas
  - Aclaris Investigational Site, San Antonio, Texas
- Bulgaria (4):
  - Aclaris Investigational Site, Pleven
  - Aclaris Investigational Site, Plovdiv
  - Aclaris Investigational Site, Sofia
  - Aclaris Investigational Site, Varna
- Czechia (6):
  - Aclaris Investigational Site, Brno
  - Aclaris Investigational Site, Hlučín
  - Aclaris Investigational Site, Ostrava
  - Aclaris Investigational Site, Pardubice
  - Aclaris Investigational Site, Prague
  - Aclaris Investigational Site, Uherské Hradiště
- Poland (20):
  - Aclaris Investigational Site, Krakow, Lesser Poland Voivodeship
  - Aclaris Investigational Site, Tomaszów Lubelski, Lubelski
  - Aclaris Investigational Site, Lublin, Lublin Voivodeship
  - Aclaris Investigational Site, Nadarzyn, Masovian Voivodeship
  - Aclaris Investigational Site, Grodzisk Mazowiecki, Mzowieckie
  - Aclaris Investigational Site, Bialystok, Podlaskie Voivodeship
  - Aclaris Investigational Site, Katowice, Silesian Voivodeship
  - Aclaris Investigational Site, Elblag, Warm.Maz.
  - Aclaris Investigational Site, Olsztyn, Warmińsko-Mazurskien
  - Aclaris Investigational Site, Poznan, Wielkopolska
  - Aclaris Investigational Site, Bialystok
  - Aclaris Investigational Site, Dąbrówka
  - Aclaris Investigational Site, Krakow
  - Aclaris Investigational Site, Lublin
  - Aclaris Investigational Site, Nowa Sól
  - Aclaris Investigational Site, Poznan
  - Aclaris Investigational Site, Sochaczew
  - Aclaris Investigational Site, Torun
  - Aclaris Investigational Site, Warsaw
  - Aclaris Investigational Site, Wroclaw